CLINICAL TRIAL: NCT05275309
Title: Determination of Optimal Positive End-expiratory Pressure Using Electrical Impedance Tomography in Children Under General Anesthesia: Comparison Between Supine and Prone Positions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H2111-072-1272
Record Dates: First submitted 2021-11-19; First posted 2022-03-11 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2021-11

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Supine Position; Prone Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children <= 1 years old (Experimental): Pediatric patients <= 1 years old of age scheduled for surgery in the prone position
  Interventions: Other: Exploration of optimal PEEP in supine and prone position

INTERVENTIONS:
Other: Exploration of optimal PEEP in supine and prone position — 1. General anesthesia is done in routine manner
  2. A sensor for electrical impedance tomography (EIT) is applied around the patient's chest.
  3. In supine position, lung recruitment maneuver is done, followed by decremental PEEP trial. Based on EIT parameter, optimal PEEP which induces minimal overdistension and collapse of lungs is determined.
  4. One hour after prone position, optimal PEEP is determined again.

SUMMARY:
The purpose of this study was to determine the appropriate positive end-expiratory pressure (PEEP) using electrical impedance tomography (EIT) in children under general anesthesia and to investigate whether there is a difference between the supine and prone positions.

ELIGIBILITY:
Inclusion Criteria:

* Children <= years of age who are scheduled for surgery in the prone position under general anesthesia

Exclusion Criteria:

* Respiratory distress, bronchopulmonary dysplasia
* Pneumothorax
* Increased intracranial pressure
* History of airway surgery
* Cervical or thoracic surgery
* Pulmonary hypertension

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Optimal PEEP level at spine position | 10 minutes after intubation (supine)
  Optimal PEEP level (cmH2O) determination using electrical impedance tomography at supine position
Optimal PEEP level at prone position | 1 hour after prone positioning (prone)
  Optimal PEEP level (cmH2O) determination using electrical impedance tomography at prone position

SECONDARY OUTCOMES:
Dynamic compliance measured using Electrical impedance tomography | until 1 hour after prone positioning
  ventilation/pressure (ml/cmH2O)
regional ventilation delay measured using Electrical impedance tomography | until 1 hour after prone positioning
  ventilation time delay during one breath (no unit)
pulmonary opening pressure measured using Electrical impedance tomography | until 1 hour after prone positioning
  alveoli opening pressure (cmH2O)
atelectasis/overdistension ratio measured using Electrical impedance tomography | until 1 hour after prone positioning
  The degree comparing atelectasis and overdistension (no unit)

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Hee-Soo Kim, Seoul, South Korea